CLINICAL TRIAL: NCT03835221
Title: Performance of Toric Hydrogel Lenses Following A Refit With Toric Silicone Hydrogel Lenses for 1 Month
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EX-MKTG-96
Record Dates: First submitted 2019-01-31; First posted 2019-02-08 (Actual); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Masking Description: Study lenses will be transferred, by an assistant, out of their packaging to unmarked new contact lens cases filled with unpreserved sterile saline just prior to dispensing to maintain subject masking of the study lenses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- methafilcon A toric / fanfilcon A toric contact lenses (Experimental): All subjects will first wear methafilcon A toric contact lenses for four (4) weeks of daily wear, then refitted with fanfilcon A toric contact lenses for four (4) weeks of daily wear.
  Interventions: Device: methafilcon A toric contact lenses; Device: fanfilcon A toric contact lenses

INTERVENTIONS:
Device: methafilcon A toric contact lenses — Bilateral daily wear of methafilcon A toric contact lenses
Device: fanfilcon A toric contact lenses — Bilateral daily wear of fanfilcon A toric contact lenses

SUMMARY:
The aim of this prospective study is to evaluate the clinical performance of habitual wearers of methafilcon A toric lenses after a refit with fanfilcon A toric lenses for 1-month of daily wear.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft contact lens wearer
* Has a contact lens spherical prescription between +6.00 to - 8.00 (inclusive)-Have no less than -0.75D of astigmatism and no more than -2.25 D in both eyes
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter
* Patient contact lens refraction should fit within the available parameters of the study lenses
* Is willing to comply with the wear schedule (at least 5 days per week, >8 hours/day assuming there are no contraindications for doing so)
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Has a Contact Lens (CL) prescription outside the range of the available parameters of the study lenses
* Has a spectacle cylinder less than -0.75D or more than -2.50 D of cylinder in either eye
* Has a history of not achieving comfortable Contact Lens (CL) wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye
* Presence of clinically significant (grade 2-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear
* Slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (past or present)
  * Seborrheic eczema, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses
* Has undergone corneal refractive surgery
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Velazquez, MSc FIACLE, Principal Investigator — School of Optometry, National Autonomous University
Locations (1):
- Optometry Clinic, National Autonomous University, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Methafilcon A / Fanfilcon A Contact Lenses: All subjects will first wear methafilcon A contact lenses for four (4) weeks of daily wear, then refitted with fanfilcon A contact lenses for four (4) weeks of daily wear.
  methafilcon A contact lenses: Bilateral daily wear of methafilcon A contact lenses
  fanfilcon A contact lenses: Bilateral daily wear of fanfilcon A contact lenses
Period: Methafilcon A
Arm/Group | Methafilcon A / Fanfilcon A Contact Lenses
Started | 43
Completed | 42
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Fanfilcon A
Arm/Group | Methafilcon A / Fanfilcon A Contact Lenses
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Lens Centration Assessment by the Investigator - Methafilcon A Toric Contact Lenses
Description: Lens centration was assessed on a 3-point scale (1=optimal centration, 2=decentration acceptable, 3=decentration unacceptable).
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Methafilcon A: All subjects will wear methafilcon A contact lenses for four (4) weeks of daily wear.
  methafilcon A contact lenses: Bilateral daily wear of methafilcon A contact lenses
Arm/Group | Methafilcon A
Number analyzed (Participants) | 43
Participants
  Optimal Centration | 40
  Decentration acceptable | 3
  Decentration unacceptable | 0

2. Primary Outcome: Number of Participants With Lens Centration Assessment by the Investigator - Methafilcon A Toric Contact Lenses
Description: as for outcome 1
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Methafilcon A
Number analyzed (Participants) | 42
Participants
  Optimal centration | 41
  Decentration acceptable | 1
  Decentration unacceptable | 0

3. Primary Outcome: Number of Participants With Lens Centration Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 1
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Fanfilcon A: All subjects will wear fanfilcon A contact lenses for four (4) weeks of daily wear.
  fanfilcon A contact lenses: Bilateral daily wear of fanfilcon A contact lenses
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
Participants
  Optimal centration | 42
  Decentration acceptable | 0
  Decentration unacceptable | 0

4. Primary Outcome: Number of Participants With Lens Centration Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 1
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
Participants
  Optimal centration | 42
  Decentration acceptable | 0
  Decentration unacceptable | 0

5. Primary Outcome: Number of Participants With Lens Centration Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 1
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
Participants
  Optimal centration | 42
  Decentration acceptable | 0
  Decentration unacceptable | 0

6. Primary Outcome: Percentage of Participants With Corneal Coverage Assessment by the Investigator - Methafilcon A Toric Contact Lenses
Description: Corneal coverage was collected on a YES/NO response. Yes - lens covers the cornea, No - lens does not cover the cornea
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Methafilcon A
Number analyzed (Participants) | 43
percentage of participants
  Yes | 100
  No | 0

7. Primary Outcome: Percentage of Participants With Corneal Coverage Assessment by the Investigator - Methafilcon A Toric Contact Lenses
Description: Corneal coverage was collected on a YES/NO response. Yes - lens covers the cornea, No - lens does not cover the cornea
Time Frame: 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Methafilcon A
Number analyzed (Participants) | 42
percentage of participants
  Yes | 100
  No | 0

8. Primary Outcome: Percentage of Participants With Corneal Coverage Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: Corneal coverage was collected on a YES/NO response. Yes - lens covers the cornea, No - lens does not cover the cornea
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
percentage of participants
  Yes | 100
  No | 0

9. Primary Outcome: Percentage of Participants With Corneal Coverage Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: Corneal coverage was collected on a YES/NO response. Yes - lens covers the cornea, No - lens does not cover the cornea
Time Frame: 2 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
percentage of participants
  Yes | 100
  No | 0

10. Primary Outcome: Percentage of Participants With Corneal Coverage Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: Corneal coverage was collected on a YES/NO response. Yes - lens covers the cornea, No - lens does not cover the cornea
Time Frame: 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
percentage of participants
  Yes | 100
  No | 0

11. Primary Outcome: Post-blink Movement Assessment by the Investigator - Methafilcon A Toric Contact Lenses
Description: Post-blink movement was assessed on a 0-4 scale (where: 0=Insufficient, unacceptable movement,1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methafilcon A
Number analyzed (Participants) | 43
units on a scale | 2.0 (0.0)

12. Primary Outcome: Post-blink Movement Assessment by the Investigator - Methafilcon A Toric Contact Lenses
Description: as for outcome 11
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methafilcon A
Number analyzed (Participants) | 42
units on a scale | 1.97 (0.15)

13. Primary Outcome: Post-blink Movement Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 11
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
units on a scale | 2.0 (0.0)

14. Primary Outcome: Post-blink Movement Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 11
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
units on a scale | 1.97 (0.15)

15. Primary Outcome: Post-blink Movement Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 11
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
units on a scale | 1.97 (0.15)

16. Primary Outcome: Lens Orientation in Primary Position of Gaze Assessment by the Investigator - Methalfilcon A Toric Contact Lenses
Description: Lens orientation was assessed in 5-degree steps with the slit lamp by measuring the amount of mislocation of the axis mark on the lens relative to the 6 o'clock position.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Methafilcon A
Number analyzed (Participants) | 43
Degrees | 2.21 (4.0)

17. Primary Outcome: Lens Orientation in Primary Position of Gaze Assessment by the Investigator - Methalfilcon A Toric Contact Lenses
Description: as for outcome 16
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Methafilcon A
Number analyzed (Participants) | 42
Degrees | 1.55 (3.2)

18. Primary Outcome: Lens Orientation in Primary Position of Gaze Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 16
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
Degrees | 0.71 (1.8)

19. Primary Outcome: Lens Orientation in Primary Position of Gaze Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 16
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
Degrees | 0.71 (1.8)

20. Primary Outcome: Lens Orientation in Primary Position of Gaze Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 16
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
Degrees | 0.47 (1.9)

21. Primary Outcome: Rotational Recovery Assessment by the Investigator - Methafilcon A Toric Contact Lenses
Description: Lens rotational recovery was assessed in 5-degree steps 1 minute after the lens was manually rotated 45degrees temporally from the primary gaze position
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Methafilcon A
Number analyzed (Participants) | 43
Degrees | 2.79 (4.8)

22. Primary Outcome: Rotational Recovery Assessment by the Investigator - Methafilcon A Toric Contact Lenses
Description: as for outcome 21
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Methafilcon A
Number analyzed (Participants) | 42
Degrees | 2.02 (3.5)

23. Primary Outcome: Rotational Recovery Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 21
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
Degrees | 0.83 (2.2)

24. Primary Outcome: Rotational Recovery Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 21
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
Degrees | 0.95 (2.3)

25. Primary Outcome: Rotational Recovery Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 21
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
Degrees | 0.48 (1.5)

26. Primary Outcome: Overall Stability Assessment by the Investigator - Methafilcon A Toric Contact Lenses
Description: Overall lens stability was assessed using a 0 - 4 scale (where 0 = very poor stability, and 4 = excellent stability).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methafilcon A
Number analyzed (Participants) | 43
units on a scale | 3.8 (0.4)

27. Primary Outcome: Overall Stability Assessment by the Investigator - Methafilcon A Toric Contact Lenses
Description: Overall lens stability was assessed using a 0 - 4 scale (where 0 = very poor stability, and 4 = excellent stability).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methafilcon A
Number analyzed (Participants) | 42
units on a scale | 3.8 (0.4)

28. Primary Outcome: Overall Stability Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: Overall lens stability was assessed using a 0 - 4 scale (where 0 = very poor stability, and 4 = excellent stability).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
units on a scale | 4.0 (0.2)

29. Primary Outcome: Overall Stability Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: Overall lens stability was assessed using a 0 - 4 scale (where 0 = very poor stability, and 4 = excellent stability).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
units on a scale | 4.0 (0.2)

30. Primary Outcome: Overall Stability Assessment by the Investigator - Fanfilcon A Toric Contact Lenses
Description: Overall lens stability was assessed using a 0 - 4 scale (where 0 = very poor stability, and 4 = excellent stability).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
units on a scale | 4.0 (0.2)

31. Primary Outcome: Overall Lens Fit Acceptance by the Investigator - Methafilcon A Toric Contact Lenses
Description: Overall lens fit acceptance assessed using grade (0-4) 0=Should not be worn, 1=Borderline but unacceptable, 2=Minimal acceptable, early review, 3=Not perfect but okay to dispense, 4=perfect.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methafilcon A
Number analyzed (Participants) | 43
units on a scale | 3.8 (0.4)

32. Primary Outcome: Overall Lens Fit Acceptance by the Investigator - Methafilcon A Toric Contact Lenses
Description: as for outcome 31
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methafilcon A
Number analyzed (Participants) | 42
units on a scale | 3.8 (0.4)

33. Primary Outcome: Overall Lens Fit Acceptance by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 31
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
units on a scale | 4.0 (0.2)

34. Primary Outcome: Overall Lens Fit Acceptance by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 31
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
units on a scale | 4.0 (0.2)

35. Primary Outcome: Overall Lens Fit Acceptance by the Investigator - Fanfilcon A Toric Contact Lenses
Description: as for outcome 31
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
units on a scale | 4.0 (0.2)

36. Secondary Outcome: Average Daily Wearing Time - Methafilcon A Toric Contact Lenses
Description: Average daily wearing time response by the subject
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours / day
Arm/Group | Methafilcon A
Number analyzed (Participants) | 42
hours / day | 10.4 (2.8)

37. Secondary Outcome: Average Daily Wearing Time - Fanfilcon A Toric Contact Lenses
Description: Average daily wearing time response by the subject
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
hours/day | 10.6 (2.8)

38. Secondary Outcome: Average Daily Wearing Time - Fanfilcon A Toric Contact Lenses
Description: Average daily wearing time response by the subject
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
hours/day | 11.0 (2.8)

39. Secondary Outcome: Average Comfortable Wearing Time - Methafilcon A Toric Contact Lenses
Description: Average comfortable wearing time - response by the subject
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Methafilcon A
Number analyzed (Participants) | 42
hours/day | 7.6 (2.8)

40. Secondary Outcome: Average Comfortable Wearing Time - Fanfilcon A Toric Contact Lenses
Description: Average comfortable wearing time - response by the subject
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
hours/day | 8.1 (2.9)

41. Secondary Outcome: Average Comfortable Wearing Time - Fanfilcon A Toric Contact Lenses
Description: Average comfortable wearing time - response by the subject
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Fanfilcon A
Number analyzed (Participants) | 42
hours/day | 8.6 (3.1)

ADVERSE EVENTS:
Time Frame: From baseline up to 8 weeks
Groups:
- Methafilcon A Toric Contact Lenses: All subjects will first wear methafilcon A toric contact lenses for four (4) weeks of daily wear, then refitted with fanfilcon A toric contact lenses for four (4) weeks of daily wear.
  methafilcon A toric contact lenses: Bilateral daily wear of methafilcon A toric contact lenses
- Fanfilcon A Toric Contact Lenses: All subjects will first wear methafilcon A toric contact lenses for four (4) weeks of daily wear, then refitted with fanfilcon A toric contact lenses for four (4) weeks of daily wear.
  fanfilcon A toric contact lenses: Bilateral daily wear of fanfilcon A toric contact lenses
Arm/Group | Methafilcon A Toric Contact Lenses | Fanfilcon A Toric Contact Lenses
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT03835221/Prot_SAP_001.pdf